CLINICAL TRIAL: NCT03628040
Title: Erector Spinae Plane Block for Video-assisted Thoracoscopic Surgery: a Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block for Video-assisted Thoracoscopic Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Cheng Lin, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112452
Record Dates: First submitted 2018-07-25; First posted 2018-08-14 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Thoracic Surgery; Peripheral Nerve Block; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: The study will be a single center (Victoria Hospital), prospective randomized, patient and assessor blinded randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization sequence will be computer-generated. Allocation concealment will be carried out via concealed assignments in opaque, sealed, and consecutively numbered envelopes. Blinding will be achieved by sham blocks. After patient allocation, a research assistant not participating in the clinical care and outcome assessment will prepare a syringe of 30 mL 0.5% ropivacaine or normal saline labeled "study drug" which will then be passed on to one of the investigators (CL or KK) who are blinded to patient allocation. Patients who are allocated to the "block" group (group B) will receive 0.5 ropivacaine with the ESPB while the "control" group (group C) will receive normal saline. In addition to ESPB, both group will receive multimodal systemic analgesia including acetaminophen, non-steroidal anti-inflammatory medication and an intravenous (IV) opioid patient-controlled analgesia (PCA) that provides IV opioids on patient-demand.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Block (Sham Comparator): Patient will receive a single shot of normal saline 20 mL injected at the erector spinae plane
  Interventions: Drug: Normal saline
- Erector Spinae Block (Active Comparator): Patient will receive a single shot of Ropivacaine Injection [Naropin] 0.5% 20 mL injected at the erector spinae plane
  Interventions: Drug: Ropivacaine Injection [Naropin]

INTERVENTIONS:
Drug: Ropivacaine Injection [Naropin] — Ropivacaine will be injected in the erector spinae plane
  Other Names: Erector spinae block
  Arms: Erector Spinae Block
Drug: Normal saline — Normal saline will be injected in the erector spinae plane
  Other Names: Sham block
  Arms: Sham Block

SUMMARY:
Video-Assisted Thoracoscopic Surgery (VATS) is a minimally invasive surgery that utilizes camera based scopes and specialized instruments through keyhole sized ports to remove lesions in the thoracic cavity. Despite reduced surgical trauma compared to the traditional thoracotomy approach, patients continued to experience moderate to severe postoperative pain. Pain medication such as opioids is commonly utilized for postoperative pain control but is associated with side effects. The use of nerve blocks, such as the recently described erector spinae plane block (ESPB) has been shown in case reports to reduce pain and thus has the potential to improve patient recovery and decrease the risk of pulmonary complication. This study aims to investigate the analgesic effect of ESPB in managing pain following VATS.

DETAILED DESCRIPTION:
VATS is a minimally invasive surgical technique to remove intrathoracic lesions. Using a camera based scope and specifically designed instruments, the surgery can be initiated with three "key-hole" sized incisions. At the end of the surgery, an incision is enlarged to allow removal of surgical specimen. Chest tubes are inserted at the end of procedure and sutured in between the ribs.

While acute pain after VATS is less than the traditional thoracotomy, patients still experience moderate amount of pain within the first 24 hours. Source of pain may be from diaphragm irritation, surgical incisions and chest tubes. Because of its origin on the chest wall, pain from VATS worsens with breathing. When pain is poorly controlled, it will lead to a shallow breathing pattern called "splinting" and this can progress to respiratory distress or failure. Given the high incidence of smoking history in this patient population, many would have presented with poor baseline respiratory function. Therefore, it is important to provide good pain control to allow deep breathing and cough to reduce respiratory complications[1][2].

Despite the smaller incisions, the incidence of chronic post-surgical pain (CPSP) after VATS is surprisingly similar to thoracotomy. The mechanism may be due to nerve compression by the trocar, an instrument inserted between the ribs to allow smooth manipulation of camera and surgical instruments in the thoracic cavity. Additionally, poorly controlled acute pain has also been postulated to lead to the development of CPSP, further emphasizing the importance of good analgesia[1].

Many regional analgesia techniques have been tried to improve postoperative analgesia. Thoracic epidural analgesia (TEA) remains the gold standard of pain control after thoracic surgery. Although it provides superior analgesia, its use is hindered by the rare but serious complication of epidural hematoma and abscess which may cause paralysis. Further, pain from VATS tends to be short-lived (less than 24 hours), making the risk to benefit ratio less ideal for TEA. An alternative to TEA is paravertebral block (PVB). Compared to TEA, it causes less hypotension and hematoma or abscess at the paravertebral space may be less consequential. Nevertheless, PVB is a deep block and is technically demanding which limits its wide adoption[3].

Erector spinae plane block (ESPB) is a novel nerve block that has been used for analgesia for surgeries of the chest and abdominal wall. Using a bony structure, the transverse process, as the end point, the block needle is very unlikely to cause injury to vital structures as is possible with TEA or PVB (for examples, the spinal cord, lungs and blood vessels). It is also technically easy to perform. ESPB has only been reported in case series but so far, no adverse events such as hypotension, hematoma or infection has been reported. ESPB has also showed promise in managing CPSP after thoracic surgery in a small case series[4].

Given its safety, ease of performance and efficacy, the study aims to study the analgesic efficacy of ESPB in addition to systemic analgesia compared to systemic analgesia alone in patients undergoing VATS. The hypothesis is that ESPB and systemic analgesia will provide better analgesia when compared to systemic analgesia alone.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Scheduled for an elective VATS
3. American Society of Anesthesiologists (ASA) physical status I to III

Exclusion Criteria:

1. Age < 18
2. BMI > 40
3. Patient refusal or inability to provide consent
4. Chronic pain conditions
5. Daily opioid use > 60 mg of oral morphine equivalents
6. Cognitive or psychiatric condition that makes it challenge to assess pain
7. Conversion to open thoracotomy
8. Allergy to any of the drugs used in this study
9. Contraindication to nerve blocks such as infection, severe coagulopathy or pre-existing neuropathy
10. Significant systemic cardiac, respiratory, hepatic or renal diseases
11. Postoperative admission to intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption in IV morphine equivalents | First postoperative 24 hour
  All source of opioid

SECONDARY OUTCOMES:
Opioid consumption in IV morphine equivalents | Second postoperative 24 hours
  All source of opioid
Area under curve of pain score | First postoperative 24 hour
  0 - 10 numeric rating scale for pain (0 minimal pain and 10 worst pain ever)
Area under curve of pain score | Second postoperative 24 hour
  0 - 10 numeric rating scale for pain (0 minimal pain and 10 worst pain ever)
Post-anesthetic recovery length of stay | up to 12 hours
  In minutes
Hospital length of stay | Up to 1 week
  in hours
Incidence of nausea | Up to 1 week
  patient reported sensation of nausea related to opioid intake
Incidence of vomiting | Up to 1 week
  nurse recorded incidence of vomiting related to opioid intake
Incidence of drowsiness | Up to 1 week
  lightheadedness, drowsiness reported by patient related to opioid intake
Incidence of pruritus | Up to 1 week
  new onset of pruritus related to opioid intake
Incidence of infection at block injection site | Up to 1 week
  defined as redness, swelling, tenderness and/or prurulent discharge
Incidence of symptomatic hematoma at block injection site | Up to 1 week
  collection of blood confirmed by ultrasound
Incidence of paresthesia in the area covered by block | Up to 1 week
  paresthesia, decreased sensation thought to related to block
Incidence of hypoxia | during the first 24 hours
  hypoxia (SaO2 < 90%) despite > 5 L oxygen
Incidence of mechanical ventilation | during the first 24 hours
  requiring re-intubation
Incidence of tachypnea | during the first 24 hours
  Respiratory rate more than 30 for more than 2 hours

IPD SHARING:
Plan to Share IPD: Undecided